CLINICAL TRIAL: NCT04495387
Title: Improving Food Pleasure and Intake of Oncology Patients Receiving Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Giandomenico Roviello, Assistant professor, md, phd, University of Florence
Other Study IDs: ALTERTASTE
Record Dates: First submitted 2020-07-23; First posted 2020-07-31 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Colon Cancer; Breast Cancer; Chemotherapeutic Toxicity
MeSH Terms: conditions — Colonic Neoplasms; Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with colon cancer
  Interventions: Drug: Chemotherapy
- patients with breast cancer
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — standard adjuvat chemotherapy for reast and colo cancer

SUMMARY:
The global cancer burden is estimated to have risen to 18.1 million new cases in 2018 (WHO), with a trend of ongoing growth. This very frequent illness exerts tremendous physical, emotional and financial strain on individuals, families, communities and health systems.

Malnutrition (under- or over-nutrition) is highly prevalent in cancer patients receiving chemotherapy and is an important predictor of morbidity, mortality, treatment response and toxicity. Alterations in taste and smell are frequently reported as side effect of chemotherapy and may contribute strongly to malnutrition and to a worsen quality of life and wellbeing social, emotional, and role functioning. There are evidences that chemotherapy influences food liking and appetite with implications for food behaviours, including food enjoyment, food preference and dietary intake. A linkage between alterations in taste and /or smell and food behaviours has been reported by some studies but not all, suggesting that there is a need for more research using common standardised methodologies and larger sample size to gain a further insight into this topic.

ELIGIBILITY:
Inclusion Criteria:

* pathological diagnosis of colorectal or breast cacer
* indication to adjuvant chemotherapy for colon cancer according local guide lines
* indication to (neo)-adjuvant chemotherapy for reast cancer according local guide lines
* possiility to sign an informed consent

Exclusion Criteria:

* patients aged <18 years
* patients aged >80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data will be collected on patients that are receiving chemotherapy for breast (n=50) and colorectal cancer (n=50) as adjuvant or neo-adjuvant therapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
change of taste chemotherapy-related alterations | the variables will be measured at four time points: before chemotherapy (T0), after 4 cycles (T1, each cycle is 21 days), at the end of chemotherapy (T2, 6 months from T0) and three months after the conclusion of the therapy (T3, 9 months from T0)
  To better understand alteration of taste/smell and food behaviours by the self-report responses, using an adapted version of a questionnaire set up to measure taste changes due to COVID-19

SECONDARY OUTCOMES:
Emotions elicited by foods | the variables will be measured at four time points: before chemotherapy (T0), after 4 cycles (T1, each cycle is 21 days), at the end of chemotherapy (T2, 6 months from T0) and three months after the conclusion of the therapy (T3, 9 months from T0)
  Emotions elicited by foods will be measured on a selection of foods through an EmoSemio questionnaire, a self-report measure of emotion developed based on preliminary interviews

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Spinelli S, Mini E, Monteleone E, Angiolini C, Roviello G. ALTERTASTE: improving food pleasure and intake of oncology patients receiving chemotherapy. Future Oncol. 2021 Jul;17(20):2573-2579. doi: 10.2217/fon-2020-0871. Epub 2021 Apr 16. PMID 33858202